CLINICAL TRIAL: NCT01596309
Title: Study of the Effect of Ready-cooked Meals Containing Cocoa Extract, as a Potential Functional Ingredient, on Cardiovascular Risk Markers in Older Population
Brief Title: Cocoa Extract-enriched Meals and Cardiovascular Risk in Older Population
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Clinica Universidad de Navarra, Universidad de Navarra (Other)
Collaborators: University of Navarra (Other)
Responsible Party: Principal Investigator, Alfredo Martinez, Professor of Nutrition and Bromatology, Clinica Universidad de Navarra, Universidad de Navarra
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: UNAV-006/2012
Record Dates: First submitted 2012-05-09; First posted 2012-05-10 (Estimated); Last update posted 2013-06-18 (Estimated); Status verified 2012-09

CONDITIONS: Cardiovascular Risk Factors
Keywords: cardiovascular risk; Elderly population; cocoa extract; overweight and obesity; Glycemic profile; lipid profile; antioxidant status; inflammatory state; Cardiovascular Risk factors in elder population
MeSH Terms: conditions — Overweight; Obesity | interventions — Chocolate; Fast Foods

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- control group, placebo (Placebo Comparator): This period will consist on a structured personalised hypocaloric diet containing ready prepared meals without extract added
  Interventions: Dietary Supplement: Cocoa extract
- Intervention group, cocoa extract (Experimental): This period will consist on a structured personalised hypocaloric diet containing ready prepared meals with cocoa extract added. Final cocoa extract daily intake will be of 1.4 g.
  Interventions: Dietary Supplement: Cocoa extract

INTERVENTIONS:
Dietary Supplement: Cocoa extract — Participants will follow a hypocaloric diet during two periods of 4 weeks, each. Within these diets, participants will consume daily 2 ready prepared frozen meals containing cocoa extract (0.7 g per meal; 1.4g per day) or nothing (placebo).
  Other Names: Ready prepared meals; bioactive ingredients

SUMMARY:
Obesity prevalence in elderly populations has increased in the last years, and the reduction of overweight and obesity is a priority target in populations of all age ranges worldwide. Obesity is a disease frequently accompanied by a pro-inflammatory state, in which metabolic functions may be compromised, and therefore there is a risk of developing comorbidities such as type-2 diabetes, hyperlipidemias, hypertension, atherosclerosis, etc. In this context, plant extracts are a good source of antioxidant compounds. Among these compounds, polyphenols have been shown to have an important antioxidant effect. Scientific evidence based on epidemiological studies suggest that flavonoids from the diet play an important role on the prevention of cardiovascular disease. Cocoa and related products are an important source of flavonoids, providing even more than tea or wine. Generally, benefits associated to cocoa consumption are related to the ability for improving lipid profile and insulin sensitivity, reducing blood pressure, platelet activity and improving endothelial dysfunction. Some studies have also shown an improvement of inflammatory conditions, mainly due to the capacity of the polyphenols contained to modify cellular transcription, and the secretion of proinflammatory cytokines in peripheral blood mononuclear cells, macrophages and lymphocytic strains. Therefore, the hypothesis of this study is that the consumption of cocoa extract-enriched prepared meals, within a hypocaloric diet, will help to reduce body weight and to improve cardiovascular risk factors compared to the same diet with standard prepared meals.

ELIGIBILITY:
Inclusion Criteria:

* Body Mass Index between 27 and 35.5 kg/m2
* Subjects with central adiposity (waist circumference over 94 cm in males and 80 cm in females)
* Subjects presenting insulin resistance non pharmacologically treated
* Subjects presenting hyperlipidemia non pharmacologically treated

Exclusion Criteria:

* Subjects following dietotherapy to loose weight at the moment of the study or in the past three months.
* Subjects with variations of weight greater than 5% of their body weight in the last three months).
* Subjects with deficient nutritional or hydration status.
* Subjects suffering from chronic diseases such as cancer, diabetes, hyperlipidemia, etc.
* Subjects with functional or structural impairments in digestive tract (peptic ulcer, malabsorption syndrome, inflammatory state, etc.)
* Subjects having gone under digestive surgery and have permanent consequences.
* Subjects suffering from allergy to cocoa or derived products.
* Subjects being physically or psychologically affected, with difficulties to attend the facilities with the required frequency.
* Smokers and frequent (more than 3 portions of beer/wine/spirits per day in males and 2 portions of beer/wine/spirits per day in females)

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2012-01; Primary Completion 2012-07 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Change from baseline of Plasma Oxidized LDL | Baseline and 4 weeks
  Levels of LDL-ox in plasma will be analysed at the beginning and the end (4 weeks) of each intervention period

SECONDARY OUTCOMES:
Change from baseline of fat mass content | Baseline and 4 weeks
  Fat mass will be measured by bioelectric impedance and Dual X-ray absorptiometry at baseline and the end (4 weeks) of each intervention period
Change from baseline of waist circumference | Baseline and 4 weeks
  Waist circumference will be measured with a measure tape at baseline and the end (4 weeks) of each intervention period
Change from baseline of hip circumference | Baseline and 4 weeks
  Hip circumference will be measured with a measure tape at baseline and the end (4 weeks) of each intervention period
Height | Baseline
Change from baseline of body weight | Baseline and 2 weeks
Change from baseline of body weight | Baseline and 4 weeks
Change from baseline of skinfolds | Baseline and 4 weeks
  Tricipital, Bicipital, subscapular and suprailiac skinfolds will be measured at baseline and the end (4 weeks) of each intervention period
Change from baseline of serum glucose levels | Baseline and 4 weeks
  Serum glucose concentration will be measured in a fasting state at the beginning and the end (4 weeks) of each intervention period
Change from baseline of serum insulin concentration | Baseline and 4 weeks
  Serum insulin concentration will be measured in a fasting state at the beginning and the end (4 weeks) of each intervention period
Change from baseline of serum free fatty acids concentration | Baseline and 4 weeks
  Serum free fatty acids concentration will be measured in a fasting state at the beginning and the end (4 weeks) of each intervention period
Change from baseline of serum total cholesterol concentration | Baseline and 4 weeks
  Serum total cholesterol concentration will be measured in a fasting state at the beginning and the end (4 weeks) of each intervention period
Change from baseline of serum HDL-cholesterol concentration | Baseline and 4 weeks
  Serum HDL-cholesterol concentration will be measured in a fasting state at the beginning and the end (4 weeks) of each intervention period
Change from baseline of serum LDL-cholesterol concentration | Baseline and 4 weeks
  Serum LDL-cholesterol concentration will be measured in a fasting state at the beginning and the end (4 weeks) of each intervention period
Change from baseline of serum triglycerides concentration | Baseline and 4 weeks
  Serum triglycerides concentration will be measured in a fasting state at the beginning and the end (4 weeks) of each intervention period
Change from baseline of serum total protein concentration | Baseline and 4 weeks
  Serum total protein concentration will be measured in a fasting state at the beginning and the end (4 weeks) of each intervention period
Change from baseline of serum transaminases concentration | Baseline and 4 weeks
  Serum transaminases (AST & ALT) concentration will be measured in a fasting state at the beginning and the end (4 weeks) of each intervention period
Change from baseline of serum homocystein concentration | Baseline and 4 weeks
  Serum homocystein concentration will be measured in a fasting state at the beginning and the end (4 weeks) of each intervention period
Change from baseline of Diastolic blood pressure | Baseline and 4 weeks
  Diastolic blood pressure will be measured at baseline and the end (4 weeks) of each intervention period
Change from baseline of Systolic blood pressure | Baseline and 4 weeks
  Systolic blood pressure will be measured at baseline and the end (4 weeks) of each intervention period
Change from baseline of Food intake | Baseline and 4 weeks
  Food intake will be measured by a 72 h weighed food record at baseline and the end (4 weeks) of each intervention period
Change from baseline of plasma PAI-1 concentration | Baseline and 4 weeks
  Plasma PAI-1 concentration will be measured in a fasting state at the beginning and the end (4 weeks) of each intervention period
Change from baseline of plasma malonyldialdehyde (MDA) concentration | Baseline and 4 weeks
  Plasma MDA concentration will be measured in a fasting state at the beginning and the end (4 weeks) of each intervention period
Change from baseline of plasma total antioxidant capacity (TAC) | Baseline and 4 weeks
  Plasma TAC will be measured in a fasting state at the beginning and the end (4 weeks) of each intervention period
Change from baseline of serum uric acid levels | Baseline and 4 weeks
  Serum uric acid levels will be measured in a fasting state at the beginning and the end (4 weeks) of each intervention period
Change from baseline of Glutathione peroxidase activity | Baseline and 4 weeks
  Glutathione peroxidase activity will be measured in a fasting state at the beginning and the end (4 weeks) of each intervention period
Change from baseline of plasma C-Reactive Protein levels | Baseline and 4 weeks
  C-Reactive Protein levels will be measured in a fasting state at the beginning and the end (4 weeks) of each intervention period
Change from baseline of plasma IL-6 levels | Baseline and 4 weeks
  IL-6 levels will be measured in a fasting state at the beginning and the end (4 weeks) of each intervention period
Change from baseline of plasma TNF-alpha levels | Baseline and 4 weeks
  TNF-alpha levels will be measured in a fasting state at the beginning and the end (4 weeks) of each intervention period
Personality Test | Baseline
  Personality will be evaluated through the NEO-PI-R test.
Change from baseline of depression degree | Baseline and 4 weeks
  Depression degree will be evaluated through the Beck depression inventory, the anxiety/STAI inventory and subjective anxiety and depression thermometer scale, at the beginning and the end of each intervention period
Change from baseline of health status | Baseline and 4 weeks
  Health status will be evaluated through the SF-36v2 Health survey at the beginning and the end of each intervention period
Change from baseline of plasma VCAM-1 levels | Baseline and 4 weeks
  VCAM-1 levels will be measured in a fasting state at the beginning and the end (4 weeks) of each intervention period
Change from baseline of plasma ICAM-1 levels | Baseline and 4 weeks
  ICAM-1 levels will be measured in a fasting state at the beginning and the end (4 weeks) of each intervention period
Cocoa Bioavailability | Baseline and 4 weeks
  Metabolites from cocoa polyphenols will be analysed in plasma and urine at the beginning and the end of each intervention period in order to estimate the bioavailability of cocoa extract studied.
DNA damage | Baseline and 4 weeks
  DNA ability to self-repair and DNA damage extent will be quantified through commet assay at the beginning and the end of each intervention period.

CONTACTS AND LOCATIONS:
Overall Officials: J. Alfredo Martinez, PhD, RN, Principal Investigator — University of Navarra, Pamplona, Spain; M. Angeles Zulet, PhD, Study Chair — University of Navarra, Pamplona, Spain; Santiago Navas-Carretero, PhD, Study Chair — University of Navarra, Pamplona, Spain; Idoia Ibero, M. Sc, Study Chair — University of Navarra, Pamplona, Spain
Locations (1):
- Department of Nutrition, Food Science, Physiology and Toxicology. University of Navarra, Pamplona, Navarre, Spain

REFERENCES:
- [Derived] Ibero-Baraibar I, Perez-Cornago A, Ramirez MJ, Martinez JA, Zulet MA. An Increase in Plasma Homovanillic Acid with Cocoa Extract Consumption Is Associated with the Alleviation of Depressive Symptoms in Overweight or Obese Adults on an Energy Restricted Diet in a Randomized Controlled Trial. J Nutr. 2015 Apr 1;146(4):897S-904S. doi: 10.3945/jn.115.222828. PMID 26962189
- [Derived] Ibero-Baraibar I, Azqueta A, Lopez de Cerain A, Martinez JA, Zulet MA. Assessment of DNA damage using comet assay in middle-aged overweight/obese subjects after following a hypocaloric diet supplemented with cocoa extract. Mutagenesis. 2015 Jan;30(1):139-46. doi: 10.1093/mutage/geu056. PMID 25527736
- [Derived] Ibero-Baraibar I, Navas-Carretero S, Abete I, Martinez JA, Zulet MA. Increases in plasma 25(OH)D levels are related to improvements in body composition and blood pressure in middle-aged subjects after a weight loss intervention: Longitudinal study. Clin Nutr. 2015 Oct;34(5):1010-7. doi: 10.1016/j.clnu.2014.11.004. Epub 2014 Nov 11. PMID 25434574
- [Derived] Ibero-Baraibar I, Abete I, Navas-Carretero S, Massis-Zaid A, Martinez JA, Zulet MA. Oxidised LDL levels decreases after the consumption of ready-to-eat meals supplemented with cocoa extract within a hypocaloric diet. Nutr Metab Cardiovasc Dis. 2014 Apr;24(4):416-22. doi: 10.1016/j.numecd.2013.09.017. Epub 2013 Nov 1. PMID 24462367